CLINICAL TRIAL: NCT05499637
Title: Pilot Study to Evaluate the Accuracy of [68Ga]Ga-PentixaFor PET/CT in the Diagnosis of Three Clinical Entities of Acute Myocardial Inflammation
Brief Title: [68Ga]Ga-PentixaFor PET/CT in Acute Myocardial Inflammation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: John O. Prior (Other)
Responsible Party: Sponsor-Investigator, John O. Prior, Head of Nuclear Medicine and Molecular Imaging Department, MD, PhD, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-00425
Record Dates: First submitted 2022-06-22; First posted 2022-08-12 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Acute Cellular Graft Rejection; Cardiac Sarcoidosis; Myocarditis Due to Drug

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- acute cellular cardiac allograft rejection (Experimental): [68Ga]Ga-PentixaFor PET/CT
  Interventions: Drug: [68Ga]Ga-PentixaFor PET/CT
- cardiac sarcoidosis (Experimental): [68Ga]Ga-PentixaFor PET/CT
  Interventions: Drug: [68Ga]Ga-PentixaFor PET/CT
- immune checkpoint inhibitor induced myocarditis (Experimental): [68Ga]Ga-PentixaFor PET/CT
  Interventions: Drug: [68Ga]Ga-PentixaFor PET/CT

INTERVENTIONS:
Drug: [68Ga]Ga-PentixaFor PET/CT — [68Ga]Ga-PentixaFor PET/CT
  Other Names: no other intervention name

SUMMARY:
Acute myocardial inflammation is an heterogenic syndrome involving different clinical pathologies with different outcome. For the purpose of this study protocol, we focuse on three entities of this syndrome, namely the acute cellular cardiac allograft rejection (ACR), cardiac sarcoidosis (CS) and the immune checkpoint inhibitor induced myocarditis (ICIM), for which non-invasive diagnosis remains challenging.

Since accurate diagnosis of myocardial inflammation in an early stage is crucial, this study aims to investigate the accuracy of [68Ga]Ga-PentixaFor as a marker of for the presence of inflammatory cells (T-lymphocytes and M1) in described patients.

The identification of a correlation between [68Ga]Ga-PentixaFor myocardial accumulation with currently accepted diagnostic tools would open up new ways to non-invasively diagnose acute myocardial inflammation.

DETAILED DESCRIPTION:
Imaging will consist of administration of maximum 50 µg IV PentixaFor, labelled with 150 ±15 MBq of 68Ga, as bolus injection 60 ±15 minutes prior PET/CT

ELIGIBILITY:
Inclusion Criteria:

* signed written informed consent
* male or female
* age ≥ 18 years
* patients with suspicion CS (group II) or ICIM (group III) or in their regular follow-up in their first year after HT (group I)
* SOC clinical follow-up at the cardiology department in CHUV.

Exclusion Criteria:

The presence of any one of the following exclusion criteria will lead to exclusion of the participant:

* absence of a signed written informed consent
* patients aged < 18 years
* claustrophobia
* myocardial ischemia in non-invasive perfusion test or coronarography in group II and III
* clinically unstable cardiovascular conditions, including:

  * clinically unstable brady-tachyarrhythmia
  * severe and symptomatic hypo- or hypertension with documented systolic blood pressure < 90 mmHg or ≥220 mmHg respectively
  * cardiogenic shock.
* women who are pregnant or breast feeding
* intention to become pregnant during the course of the study in group II
* previous enrolment into the current study
* moderate to severe renal insufficiency (GFR < 45 mL/min/1,73 m2), with contra-indication to the administration of Gadolinium in group II and III
* enrollment of the investigator, his/her family members, employees and other dependent persons
* history of any disease or relevant physical or psychiatric condition or abnormal physical finding which may interfere with the study objectives at the investigator judgment
* insufficient knowledge of project language, inability to give consent or to follow procedures
* the patient makes use of his/her "right not to know" and refuses to be informed about incidental findings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Imaging results obtained by [68Ga]Ga-PentixaFor PET/CT - lesion number | 1 year
  lesion number imaged
Imaging results obtained by [68Ga]Ga-PentixaFor PET/CT - lesion site | 1 year
  lesion sites imaged
Imaging results obtained by [68Ga]Ga-PentixaFor PET/CT - SUV | 1 year
  standard uptake value

SECONDARY OUTCOMES:
to assess toxicity data | 1 year
  analysis of collected AEs classified according to CTCAE version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: John O Prior, MD, PhD, Study Chair — University of Lausanne Hospitals
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No